CLINICAL TRIAL: NCT03895073
Title: Observation Study for the Assessment of the "Four-point" Questionnaire by Severo and His Associates and Its Weighting in the Greek Population to Provide a Powerful Tool for Categorizing the Severity of the Symptoms of Heart Failure
Brief Title: HEart fAiluRe evaluaTion Questionnaire
Acronym: HEART
Status: Completed | Type: Observational
Sponsor: John Parissis (Other)
Responsible Party: Sponsor-Investigator, John Parissis, Associate Professor, Attikon Hospital
Organization: Attikon Hospital (Other)
Other Study IDs: IIS-HEART-2018
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure; Heart Failure NYHA Class III; Heart Failure NYHA Class II; Heart Failure NYHA Class I; Heart Failure NYHA Class IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy: healthy volunteers' replies to questionnaire
  Interventions: Other: healthy volunteers
- heart failure: heart failure patients' replies the questionnaire
  Interventions: Other: healthy volunteers

INTERVENTIONS:
Other: healthy volunteers — the questionnaire has been assessed by both groups, healthy and heart failure
  Other Names: healthy vs heart failure

SUMMARY:
The "four-point" questionnaire by Severo and his associates was weighted in 2011 in the Portuguese population and aims to characterize the severity of the symptoms of heart failure by providing a way to minimize the reliability of the NYHA classification. The questionnaire consists of four closed questions, three possible single-choice answers, coded 0, 1 or 2, and has been translated into Greek in accordance with the internationally-based methodology, with forward-backward translation.

DETAILED DESCRIPTION:
In clinical practice, the most commonly used classifications of the severity of CA⸱ are the New York Heart Association functional classification (NYHA), which is based on symptoms and exercise capacity11 and has been used in the majority of clinical trials combined with the fraction left ventricular ejection and ACC / AHA (American College of Cardiology Foundation / American Heart Association), which describes the disease according to structural lesions and symptoms.

With NYHA calibration, patients can be classified into four classes (I, II, III, IV) according to conclusions drawn from the medical history and / or observations of their physical activity and in some cases from cardiac function measurements . An attempt has been made to increase the objectivity of the method through a more comprehensive assessment, which will also be based on clinical measurements from electrocardiograms, stress tests, x-rays, echocardiograms, etc. There is a very high variability among clinicians' ratings on classifying patients in classes based on the NYHA functional classification as the class is selected according to the physician's personal assessment of the patient's physical condition. This increases the subjectivity of the particular sorting system. Studies have shown that there is agreement on NYHA calibration between different doctors for the same patient, of 55%, which leads to the conclusion that the use of this scale as the endpoint in clinical research is questionable and inadequate.

Patient self-assessments are more reliable with respect to the subjectivity of assessing the severity of symptoms. This is why maximizing the interest of the scientific community, clinicians and pharmaceutical companies in developing more subjective methods of measuring health status. 30% of all new drugs developed use patient-reported outcomes (PROs) as primary or intermediate endpoints.

The different data collection methods and sampling techniques are methods and methodologies that allow for the reduction of the amount of data to be collected, considering data only as some elements of a subset of the cases under consideration. The questionnaire is a form that includes a series of structured questions, in which the respondent is asked to respond in writing and in a specific order. Questionnaires collect data asking people to answer exactly the same set of questions. They are usually used in a research strategy to collect descriptive and explanatory data about views, behaviors, features, attitudes, etc. The questionnaire is the means of communication between the researcher and the respondents, directly or indirectly, depending on the method of data collection. The structure of the questionnaire, due to its qualities, is the most critical and delicate task, crucial to the success of a statistical survey.

ELIGIBILITY:
Inclusion Criteria:

* NYHA classification
* informed consent
* compliant with study procedures

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure patients vs Healthy matched controls
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
questionnaire replies | 1 day
  rating in Severo questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John Parissis, MD, Study Chair — Attikon Hospital
Locations (1):
- Attikon Hospital, Athens, Attica, Greece